CLINICAL TRIAL: NCT00635284
Title: A Phase I Trial of ABI-009 (Nab-rapamycin) Administered Weekly in Patients With Advanced Non-hematologic Malignancies
Brief Title: ABI-009 Trial in Patients With Advanced Non-hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA401; NCT00573677 (obsolete NCT alias)
Record Dates: First submitted 2008-03-07; First posted 2008-03-13 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABI-009 (Experimental)
  Interventions: Drug: ABI-009

INTERVENTIONS:
Drug: ABI-009 — nab-rapamycin
  Other Names: nab-rapamycin

SUMMARY:
To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) of ABI-009 given weekly; to characterize the toxicities of ABI-009; and to determine the pharmacokinetic parameters for ABI-009 when given on a weekly schedule.

DETAILED DESCRIPTION:
No extended description necessary

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria to be enrolled in this study.

1. Male and female patients with histologically or cytologically confirmed diagnosis of cancer which is not amenable to curative therapy.
2. Patients with advanced non-hematologic malignancies for whom no standard therapy exists.
3. Measurable disease by RECIST or evaluable disease (e.g., bone metastasis, pleural effusion, ascites, or lesions which do not fulfill RECIST criteria for metastatic disease)
4. Off all therapy (inclusive of investigational therapies) for at least 4 weeks prior to study drug administration OR off all daily or weekly therapy (inclusive of investigational therapies) for at least 2 weeks prior to study drug administration and without any side effects associated with these therapies.
5. Female patients of child-bearing potential must have a negative serum pregnancy test within 7 days prior to first study drug administration.
6. Female patients who are postmenopausal must have 12 months of amenorrhea, surgically sterile, or must agree to the use of a physical method of non-hormonal contraception.
7. Male patients must be surgically sterile or agree to the use of a barrier method of contraception.
8. Life expectancy of > 3 months.
9. ECOG Performance Status of 0-1.
10. Patients must be able to provide informed consent indicating knowledge of his/her disease process, the investigational nature of the therapy, alternatives, benefits, and risks including potential side effects.
11. Age ≥ 18 years of age.
12. No major surgery within 4 weeks before treatment with ABI-009. (A biopsy is not considered major surgery).
13. No chemotherapy, hormonal therapy, immunotherapy or radiotherapy within 4 weeks before treatment with ABI-009 (6 weeks for previous treatment with nitrosoureas, mitomycin, or extensive radiotherapy) and no immunosuppressive agents within 3 weeks before study entry (except corticosteroids used as antiemetics).
14. No immunosuppressive agents within 3 weeks before study entry (except corticosteroids used as antiemetics).
15. Required Initial Laboratory Data:

    * Hemoglobin > 9.0 g/dL
    * WBC ≥ 3,000/µl
    * ANC ≥ 1,500/µl
    * Platelet count ≥ 100,000/µl
    * Total Bilirubin ≤ ULN
    * SGOT (AST) SGPT (ALT) ≤ 1.5 x ULN ≤ 1.5 x ULN
    * Serum Cholesterol < 350 mg/dL
    * Serum Triglyceride < 300 mg/dL
16. Adequate renal function with serum creatinine < 1.5 mg/dL and/or creatinine clearance (cockroft formula) ≥ 60 mL/min.
17. No active alcohol abuse, drug addiction, or psychotic disorders.
18. No known concomitant genetic or acquired immunosuppressive diseases (such as AIDS).
19. If obese, a patient must be treated with doses calculated using his/her actual BSA (The physician must be comfortable treating at the full BSA dose regardless of BSA).

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study.

1. Pregnant or nursing women.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition including macrolide (e.g. azithromycin, clarithromycin, dirithromycin, and erythromycin) and ketolide antibiotics.
3. Patients have not recovered from adverse affects of radiation therapy or investigational agent within previous 28 days.
4. Uncontrolled intercurrent illness that in the opinion of the investigator would limit compliance and tolerance to study requirements
5. Patients with known brain metastases or leptomeningeal tumor involvement.
6. Receiving any of the following: concomitant antitumor therapy or inhibitors of CYP3A4.
7. Patients with history of interstitial lung disease and/or pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2011-06-01 (Actual); Study Completion 2011-06-01 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) of ABI-009 administered weekly and pharmacokinetic parameters for ABI-009. | End of Study (EOS) and Follow Up

SECONDARY OUTCOMES:
Efficacy of ABI-009 in this patient population | End of Study (EOS) and Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: Ana M. Gonzalez, MD, Principal Investigator — M.D. Anderson Cancer Center; Sant P. Chawla, MD, Principal Investigator — Sarcoma Oncology Center
Locations (2):
- United States (2):
  - Sarcoma Oncology Center, Santa Monica, California
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Gonzalez-Angulo AM, Meric-Bernstam F, Chawla S, Falchook G, Hong D, Akcakanat A, Chen H, Naing A, Fu S, Wheler J, Moulder S, Helgason T, Li S, Elias I, Desai N, Kurzrock R. Weekly nab-Rapamycin in patients with advanced nonhematologic malignancies: final results of a phase I trial. Clin Cancer Res. 2013 Oct 1;19(19):5474-84. doi: 10.1158/1078-0432.CCR-12-3110. PMID 24089446